CLINICAL TRIAL: NCT03359993
Title: Umbilical Vein Needle Catheterization for Endotracheal Intubation.
Acronym: Intubation
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0417
Record Dates: First submitted 2017-11-28; First posted 2017-12-02 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-01

CONDITIONS: Infant Respiratory Distress Syndrome
Keywords: Endotracheal intubation; Neonatal premedication; Delivery room
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants intubated: All participants were preterm infants intubated in the delivery room for Infantile Respiratory Distress Syndrome (IRDS). The purpose of this research is to determine a premedication of intubation. This consists of describing a simple and effective method for premedication in the delivery room, using the umbilical vein, directly perforated through the Wharton jelly.
  Interventions: Procedure: Premedication of intubation

INTERVENTIONS:
Procedure: Premedication of intubation — The umbilical vein is punctured to inject drugs efficiently. The access is simple, the umbilical vein is clearly visible, and a blood reflux can be found easily. We used the same equipment required for a peripheral venous injection: 24 gauge cannula, antisepsis, compress, and a syringe with the prepared anesthetic drugs. We report 5 cases of intubations in the delivery room using this method to administer the premedication.

SUMMARY:
The investigators describe a simple and efficient method to give a premedication in the delivery room, using the umbilical vein, directly punctured through Wharton's jelly.

DETAILED DESCRIPTION:
The umbilical vein is punctured to inject drugs efficiently. The access is simple, the umbilical vein is clearly visible, and a blood reflux can be found easily. The investigators used the same equipment required for a peripheral venous injection: 24 gauge cannula, antisepsis, compress, and a syringe with the prepared anesthetic drugs. The investigators report 5 cases of intubations in the delivery room using this method to administer the premedication.

ELIGIBILITY:
Inclusion Criteria:

* All the patients were preterm neonates intubated in the delivery room for infant respiratory distress syndrome (IRDS).

Exclusion Criteria:

* Refusal of legal owners

Max Age: 30 Minutes | Sex: All
Age Groups: Child
Study Population: The patients were preterm neonates intubated in the delivery room for infant respiratory distress syndrome (IRDS)
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Conditions of intubation | Seven months
  Classified from bad to excellent, depending on the neonates' residual tone, vocal chords mobility, and persistence of movements while inserting the tube.

SECONDARY OUTCOMES:
Duration of intubation | Seven months
  The investigators measure the time in seconds between insertion of the tube and the end of fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne BORRHOMEE, Principal Investigator — Hôpital NOVO
Locations (1):
- Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No